CLINICAL TRIAL: NCT05945472
Title: Mental Beauty, the Unexplored Impact of Cosmetics on Mood, Personal Self-esteem, Perceived Stress, Mindfulness and Psychological Well-being.
Brief Title: Beauty as a State of Wellness Beauty as a State of Wellbeing in Women 40 to 64 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: BIT BEAUTY SL. (Unknown)
Responsible Party: Principal Investigator, Yolanda Marcen Roman, Clinical Professor, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Beauty and wellness
Record Dates: First submitted 2023-01-11; First posted 2023-07-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Self Esteem; Psychological Well-being; Stress, Physiological; Mood
Keywords: beauty; Wellness; cosmetics; self-esteem; stress; Mental Beauty
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: There are three arms, two of intervention and one control. Arm 1: intervention with fasting method Arm 2: Non-fasting method Arm 3: Control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Once participants have signed the informed consent form and meet the inclusion requirements, they are randomly assigned 1/1 to the fasting or non-fasting intervention group.
  The statistician does not know to which group the participants belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive reinforcement method (Experimental): The people who form the intervention groups will receive a facial cosmetic of natural components to be administered for 28 days, for which they will be given the cream.
  The cream will be provided to the participants on the 1st day of the talk. The container containing the facial cosmetic will be applied twice a day, morning and evening.
  Afterwards, in the "experimental" group, the participants will be given a talk on how to administer it according to the "positive reinforcement" method.
  Interventions: Other: Positive reinforcement method
- Standard method (Active Comparator): The people who form the intervention groups will receive a facial cosmetic of natural components to be administered for 28 days, for which they will be given the cream.
  The cream will be provided to the participants on the 1st day of the talk. The container containing the facial cosmetic will be applied twice a day, morning and evening.
  Interventions: Other: Standard method
- Control (No Intervention): This group will continue to use their usual cosmetics and complete the questionnaire on the first day of the study and on the last day of the study (28 days later).

INTERVENTIONS:
Other: Positive reinforcement method — A 30-minute talk based on mindfulness, positive thinking and teaching for the application of the cosmetic through positive messages (Ayuna method). Adapts the teachings of mindfulness to the field of beauty and stimulates the skin-brain connection through self-care. By applying cosmetics through intentional massages, with this technique is stimulated the brain in a positive positively in the general wellbeing.
  The cosmetic is applied with a massage aimed at loving oneself, a ceremony for the skin and an invitation to enjoy the moment; positive messages are included during the application. In addition to favoring the penetration of the products, these maneuvers help to disconnect and achieve, in the long term, a healthier appearance. The technique consists of slow, intentional movements to create an ideal space to become aware of the present moment and draw a love story with oneself.
  Arms: Positive reinforcement method
Other: Standard method — A 30-minute talk based on how to administer it according to the guidelines of general cosmetology, related to the use and application of the cream, following conventional techniques of the cosmetic industry, which focus on the application of the product in the areas of wrinkles or with more treatment needs: "anti-aging" "anti-stain" "anti-sagging" "anti-sagging" product, "anti-sagging" "anti-sagging" "anti-sagging" "anti-sagging" "anti-sagging" "anti-sagging" product. rejuvenating results to try to reduce the "skin years", reduce wrinkles, loss of firmness, flaccidity and spots.
  Arms: Standard method

SUMMARY:
The sociocultural pressure towards women's body image is one of the problems that today afflicts much of the female population. It is a reality that society exerts a strong pressure on body image, particularly on women.

The main objective of this study is to analyze the self-perception and self-esteem of people who apply a facial cosmetic. A convenience sample of 150 participants is estimated, who can be randomly included in one of the three groups with different interventions.

DETAILED DESCRIPTION:
The aging process is something inherent in all people, causing biological and structural changes in our organism, being the skin the one that shows the first signs of this aging. Being healthy is no longer a desire and a natural aspiration of every person, but a kind of tyranny that has turned health into a duty that, according to the wellness industry, can only be satisfied through the consumption of certain commercial products and services. The cosmetic industry feeds us with false beliefs where perfection is something achievable, but many women do not want false promises from the cosmetic industry when they are aware that they have wrinkles. Such practices jeopardize physical health and impact mental health.

IIn line with this evolution, the researchers propose this study that suggests a relationship between the use of cosmetics, psychological well-being, stress and self-esteem of the people who consume them.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 and 65 years old
* Who use a facial cosmetic at least once a week.

Exclusion Criteria:

* Receiving oncological treatment at the time of participation in the study.
* Suffering acute infectious disease processes in the 3 months prior to the study or during the study period.
* Being diagnosed with some type of mental illness.
* Failure to sign the informed consent form.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | 3 minutes
  The Rosenberg self-esteem scale is a test with good psychometric properties, and is one of the most widely used tests for the evaluation of self-esteem in clinical practice and scientific research. The Rosenberg Self-Esteem Scale (RSES) is made up of 10 items that refer to self-respect and self-acceptance rated on a 4-point Likert-type scale, ranging from 1 (totally disagree) to 4 (totally agree). Items 1, 3, 4, 7, and 10 are positively worded, and items 2, 5, 6, 8, and 9 negatively. Each dimension is made up of 6 items that are rated on a 99-point scale ranging from 1 (totally disagree with the item) to 99 (totally agree with the item). The higher the score, the higher the self-esteem.
Perceived Stress Scale | 5 minutes
  The "Perceived Stress Scale" (PSS), constructed in its original version, has been the instrument most frequently used to study the relationship between stress and psychological health, The questions refer to feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale ranging from 0 'never' to 4 'very often'.
  To calculate a total PSS score, the responses to the four positively stated items (items 4, 5, 7, and 8) must first be reversed (i.e., 0 => 4; 1 => 3; 2 => 2; 3 => 1 ; 4 => 0).
  Then the PSS score is obtained by adding all the elements. Higher scores indicate higher levels of perceived stress.
The Short Mood Introspection Scale | 5 minutes
  The Short Mood Introspection Scale. The scale consists of 16 adjectives that measure the mood of the current moment. Participants rate themselves on a four-point response scale (1 does not describe my mood at all, 2 describes my mood a little, 3 describes my mood well, 4 describes my mood very well). The higher the score, the greater the perception of mood.
Psychological Well-Being Scale | 10 minutes
  Ryff (Psychological Well-Being Scale). It is made up of six dimensions: Self-acceptance, positive relationships, autonomy, mastery of the environment, purpose in life, personal growth. Scale made up of 39 items to which the participants responded using a Likert-type response format with sensitive sensors between 1 (totally disagree) and 6 (totally agree), for a maximum total of 234 points. Scores above 176 are indicative of elevated psychological well-being (BP); between 141 and 175 BP high; between 117 and 140 moderate BP points; and less than 116 BP points low.
Descriptive questionnaire | 5 minutes
  Age, marital status, highest level of education, work, are you a health worker, do you work in the beauty and esthetics industry, level of income within the family unit.
  Do you currently make use of regular facial treatment, at what age did you start using cosmetics for facial use, how many years have you been using facial cosmetics, when you buy your facial treatment cosmetics what do you take into account at the time of purchase, how do you feel if you think about your body, how do you feel if you think about your face, how do you feel if you think about your body, how do you feel if you think about your face, how do you feel if you think about your body, how do you feel if you think about your body, how do you feel if you think about your face?

SECONDARY OUTCOMES:
The abbreviated 5-factor mindfulness instrument FFMQ | 10 minutes
  The abbreviated 5-factor mindfulness instrument. The FFMQ is a self-report test made up of 39 items, which measures the general tendency to proceed with Mindfulness based on five skills: Observation, Description, Acting Consciously, Absence of Judgment and Absence of Reactivity.
  There are two patterns of scoring involved in the Five Facet Mindfulness Test:
  Direct Scoring - where the items are scored according to the Likert value (for example 1 would add a score of 1 and 4 adds a value of 4).
  Reverse Scoring - where we score the items backward (for example, 1 adds a score of 5, 5 adds a score of 1, 4 would mean a score of 2, and likewise).
  Summation of all the direct and reverse items adds up to the total value of the scale.
  The responses on the scale are made on a 5-point Likert scale, and the sum of the forward and reverse scoring items gives the total score.
  The five subscales of the test provide a meaningful estimate of how aware the respondent is at the moment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. Zaragoza's University, Zaragoza, Spain

REFERENCES:
- [Background] Danthinne ES, Giorgianni FE, Austin SB, Rodgers RF. Beauty and the big business: A qualitative investigation of the development and implementation of the CVS Beauty Mark. Body Image. 2022 Jun;41:74-83. doi: 10.1016/j.bodyim.2022.01.012. Epub 2022 Feb 28. PMID 35240392
- [Background] Díaz Rojo, J. A., Y Morant Marco, R. (2007). El discurso crítico contra la <tiranía> del culto al cuerpo. Revista electrónica de estudios filológicos, (XIV), 1.
- [Background] McLaren, L. Hardy, R. Y Gauvin, L. (2004). Positive and negative body-related comments and their relationship with body dissatisfaction in middle-aged women. Psychology & health ,2, 261-272.
- [Background] Voegeli R, Schoop R, Prestat-Marquis E, Rawlings AV, Shackelford TK, Fink B. Cross-cultural perception of female facial appearance: A multi-ethnic and multi-centre study. PLoS One. 2021 Jan 22;16(1):e0245998. doi: 10.1371/journal.pone.0245998. eCollection 2021. PMID 33481957
- [Background] Little AC, Jones BC, DeBruine LM. Facial attractiveness: evolutionary based research. Philos Trans R Soc Lond B Biol Sci. 2011 Jun 12;366(1571):1638-59. doi: 10.1098/rstb.2010.0404. PMID 21536551
- [Background] Samson N, Fink B, Matts PJ. Visible skin condition and perception of human facial appearance. Int J Cosmet Sci. 2010 Jun;32(3):167-84. doi: 10.1111/j.1468-2494.2009.00535.x. Epub 2009 Nov 3. PMID 19889046
- [Background] Fares K, Hallit S, Haddad C, Akel M, Khachan T, Obeid S. Relationship Between Cosmetics Use, Self-Esteem, and Self-Perceived Attractiveness Among Lebanese Women. J Cosmet Sci. 2019 Jan/Feb;70(1):47-56. PMID 30856095
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417